CLINICAL TRIAL: NCT02145663
Title: Helsinki Ultra-acute Stroke Biomarker Study
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: HUS area Prehospital Emergency Service (Unknown)
Responsible Party: Principal Investigator, Perttu Lindsberg, Professor, Helsinki University Central Hospital
Other Study IDs: HUSBS2013; MNEURT ISCHEMIC STROKE 813 (Other: HUCH)
Record Dates: First submitted 2014-05-02; First posted 2014-05-23 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Serum and Plasma

SUMMARY:
The aim of this study is to establish diagnostic and predictive biomarkers for patients with suspected acute stroke, that are transported by EMS as candidates for thrombolytic treatment. The study focuses on the ultra acute phase, <4.5 hours from symptom onset, including the prehospital setting. Analyses will include known biomarkers (e.g. GFAP, NR2 peptide) and a discovery phase for novel markers. Patient outcome will be evaluated at 3 month using the modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke suspected by EMS personnel
* Transport to tertiary hospital as possible candidate for thrombolytic treatment of ischemic stroke
* Age ≥18
* Successful prehospital blood sampling by EMS personnel

Exclusion Criteria:

* Unsuccessful prehospital blood sampling by EMS personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected acute stroke, being transported by emergency medical services (EMS) to a tertiary hospital stroke center, as candidates for thrombolytic treatment of acute ischemic stroke.
Sampling Method: Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of biomarkers for identifying ischemic stroke, transient ischemic attack, intracerebral hemorrhage and stroke mimics. | 90 days +/- 5 days
  Metrics: Receiver operating characteristic curve analysis, sensitivity, specificity, positive predictive value, negative predictive value
Predictive accuracy of biomarkers for identifying patients not responding to thrombolytic treatment. | 90 days +/- 5 days
  Metrics: Receiver operating characteristic curve analysis, sensitivity, specificity, positive predictive value, negative predictive value
Predictive accuracy of biomarkers for identifying patients facing hemorrhagic complications of thrombolytic treatment | 90 days +/- 5 days
  Metrics: Receiver operating characteristic curve analysis, sensitivity, specificity, positive predictive value, negative predictive value
Predictive accuracy of biomarkers for predicting outcome | 90 days +/- 5 days
  Metrics: Receiver operating characteristic curve analysis, sensitivity, specificity, positive predictive value, negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Perttu Lindsberg, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Derived] Mattila OS, Puolakka T, Ritvonen J, Pihlasviita S, Harve H, Alanen A, Sibolt G, Curtze S, Strbian D, Pystynen M, Tatlisumak T, Kuisma M, Lindsberg PJ. Targets for improving dispatcher identification of acute stroke. Int J Stroke. 2019 Jun;14(4):409-416. doi: 10.1177/1747493019830315. Epub 2019 Feb 13. PMID 30758276